CLINICAL TRIAL: NCT04365738
Title: Pulmonary Rehabilitation in Post-Acute Period of COVID-19 Infection: Prospective Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation in Post-Acute Period of COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Assoc.Prof., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR COVID-19
Record Dates: First submitted 2020-04-26; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Pulmonary Rehabilitation; Dyspnea; Fatigue; Pain; Anxiety
MeSH Terms: conditions — COVID-19; Dyspnea; Fatigue; Pain; Anxiety Disorders | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation (Experimental): The patients who applied pulmonary rehabilitation were checked, motivated and followed-up regularly with video calls every day. Pulmonary rehabilitation program consists of patient education, breathing, in-house mobilization and range of motion exercises.
  Interventions: Other: Rehabilitation
- Control (Placebo Comparator): As a patient education, information was given about the disease and treatment process, listening to the patient during this process and getting regular sleep, balanced nutrition and taking a break from smokers.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Chest and diaphragm respiration, in-house mobilization, joint range of motion exercises was performed to the patients as breathing exercises.

SUMMARY:
The aim of this study is to investigate the efficacy of pulmonary rehabilitation(PR) applied in the isolation processes of post-acute patients with mild and moderate symptoms who had positive COVID-19 test on dyspnea,muscle pain,chest expansion,lower limb muscle strength and dynamic balance,fatigue,anxiety and depression.

DETAILED DESCRIPTION:
This study was conducted with 270 patients who were the COVID-19 test was positive and isolated in their homes during post-acute periods.While one of the groups (n=135) was asked to remain isolated at home by providing patient education,a PR program was applied for 4 weeks in addition to the patients in the other group(n=135).PR consists of patient education, breathing, in-house mobilization and range of motion exercises.As the evaluation parameters,pre-treatment and post-treatment dyspnea levels with Borg scale,muscle pain with visual analog scale(VAS),functional capacities with sit-up test,chest expansions with tape measure,respiratory frequency,fatigue level with fatigue severity scale,and emotional status with hospital anxiety and depression(HAD) scale were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 28-45, positive COVID-19 test, being in the post-acute period, having symptoms of mild-moderate severity, respiratory rate ≤40 breaths / min, patients who can make video speech

Exclusion Criteria:

* Severe symptom involvement, fever more than 38 degrees, obese patients, patients with multiple comorbidities, patients with one or more organ failure, oxygen saturation in the blood ≤95%, a resting blood pressure of <90/60 mmHg or> 140 / 90 mmHg patients

Ages: 28 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Dyspnea | Baseline, up to 4 weeks
  The Borg scale is a scale scored between 0-10, indicating the severity of dyspnea. 0 indicates no shortness of breath, 10 indicates severe shortness of breath

SECONDARY OUTCOMES:
Chest expansion | Baseline, up to 4 weeks
  Chest expansion was evaluated by measuring the difference between the maximum inspiration and maximum expiration from the level of xsphoid processus of the patients.
Fatigue severity | Baseline, up to 4 weeks
  Fatigue severity scale is a questionnaire consisting of 9 questions showing the degree of fatigue of patients. An average score of less than 2.8 indicates no fatigue, and more than 6.1 indicates chronic fatigue syndrome
Visual Analog Scale for pain | Baseline, up to 4 weeks
  Patients were instructed and asked to give a score between 0-10 with 0 equating to no pain, 10 indicating severe pain
Hospital anxiety and depression scale | Baseline, up to 4 weeks
  The HAD scale is a short self administered questionnaire used to screen for anxiety and depression. The questionnaire consists of 14 items, seven each measuring anxiety and seven to measure depression. According to research literature, the cut-off point for elevated anxiety and depression as measured by the HAD scale is eight

CONTACTS AND LOCATIONS:
Overall Officials: Tomri̇s Duymaz, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided